CLINICAL TRIAL: NCT01790958
Title: An Observational, Multi-Center Phase 1 Study of the Safety and Effectiveness of Frequency Specific Microcurrent Stimulation as an Alternative Treatment for Retinal Diseases
Brief Title: Microcurrent Stimulation to Treat Macular Degeneration
Status: Completed | Type: Observational
Sponsor: Retina Institute of Hawaii (Other)
Responsible Party: Sponsor
Other Study IDs: RIH 1009
Record Dates: First submitted 2013-02-11; First posted 2013-02-13 (Estimated); Last update posted 2013-02-13 (Estimated); Status verified 2013-02

CONDITIONS: Retinal Diseases; Stargardt's Disease; Retinitis Pigmentosa
MeSH Terms: conditions — Retinal Diseases; Stargardt Disease; Retinitis Pigmentosa

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Microcurrent stimulation thereapy improves retinal efficiency and may restore and/or improve retinal function.

DETAILED DESCRIPTION:
This is an observational study in which data will be collected from a group of patients with retinal diseases such as Dry Macular Degeneration, RetinitisPigmentosa, and Stargardt's Disease, who have opted to receive Microcurrent Stimulation Therapy as an alternative treatment for their retinal condition.

ELIGIBILITY:
Inclusion Criteria:

* Ability to provide written consent and comply with follow up visits
* Age 40 years or older
* ETDRS best corrected visual acuity better than 5 letters
* History of Dry Age Relted Macular Degeneration; Retinitis Pigmentosa; Stargardt's disease
* No Anti-VEGF treatments for at least 3 months prior to study
* No new antioxidant/vitamin supplementation for at least 3 months prior to study

Exclusion Criteria:

* History of Non-Compliance with regular medical visits
* Significant media opacities (exclude NS 4+) that may interfere with assessing visual acuity
* Presence of pigment epithelial tears or rips
* Known serious allergies to fluorescein dye
* Presence of retinal neovascularization
* Any treatment with an investigation agent in the past 30 days

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with retinal disease such as Age-Related Macular Degeneration, STargardt's Disease, and Retinitis Pigmentosa
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2012-06; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Measure visual acuity after receiving microcurrent stimulation treatments. | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: George Papastergiou, MD, Principal Investigator — Retina Institute of Hawaii
Locations (4):
- United States (4):
  - Hawaii Cataract Laser Institute - Hilo, Hilo, Hawaii
  - Retina Institute of Hawaii, Honolulu, Hawaii
  - Hawaii Cataract Laser Institute - Maui, Kahului, Hawaii
  - Hawaii Cataract Laser Institute - Kona, Kailua-Kona, Hawaii